CLINICAL TRIAL: NCT06363071
Title: Gait-initiation Related APA Training in Individuals With Parkinson Disease -Explicit Training and Paired Associative Stimulation(PAS) Priming
Brief Title: APA and PAS Training for Gait Initiation in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000495A3
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Gait Initiation; Balance training; Anticipatory postural adjustments; Paired associative stimulation (PAS); Transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stage 1:Healthy people (Experimental): To establish PAS baseline and reliability.
  Interventions: Procedure: Paired associative stimulation
- Stage 2:PD people (Experimental): To establish stage 3 training protocol.
  Interventions: Procedure: Paired associative stimulation
- Stage 3:PD people (No Intervention): Control group.
- Stage 3: PD APA training group (Experimental): Weight shift training and APA feedback.
  Interventions: Other: Weight shift training and APA feedback
- Stage 3:PD PAS group (Experimental): Using PAS to regulate brain plasticity
  Interventions: Procedure: Paired associative stimulation

INTERVENTIONS:
Other: Weight shift training and APA feedback — Use COP trajectory to train weight shift on force plate. To give APA visual feedback for subjects after weight shift training.
  Other Names: • APA training group
  Arms: Stage 3: PD APA training group
Procedure: Paired associative stimulation — Use TMS combine ES to stimulate TA nerve and M1 cortical
  Other Names: PAS group
  Arms: Stage 1:Healthy people; Stage 2:PD people; Stage 3:PD PAS group

SUMMARY:
Our research focused on understanding the interplay between brain excitability and balance function in patients with Parkinson's disease (PD), alongside evaluating effective physical therapy methods. It highlights the prevalence of non-motor disorders and cognitive impairments among PD patients, including balance and postural issues, cognitive function decline, and gait instability. Additionally, it notes that PD patients exhibit abnormal electrophysiological responses, indicating altered central excitability.

DETAILED DESCRIPTION:
Research on Brain Excitability and Balance Function Performance in Patients with Parkinson's Disease and Related Physical Therapy Methods

Research indicates that non-motor disorders and cognitive impairments are prevalent in most patients with Parkinson's disease. These include balance issues, postural instability, impaired cognitive functions like working memory and executive functions, and gait instability. Additionally, electrophysiological phenomena in Parkinson's disease patients reveal abnormal central excitatory and inhibitory responses compared to healthy individuals.

This experiment seeks to investigate the link between motor performance and brain excitability in patients with Parkinson's disease. Previous studies suggest that associative electrical stimulation, used to regulate sensorimotor information integration, can enhance brain excitability in both healthy individuals and those with Parkinson's disease. However, the optimal parameters for this stimulation remain uncertain.

Furthermore, balance exercise training can improve motor performance in Parkinson's disease patients. This study aims to determine if various designs of associative electrical stimulation parameters can help these patients achieve optimal brain excitability regulation. The combined approach of this stimulation and balance exercise training aims to maintain and improve the patients' functional performance, thereby enhancing the safety of their daily activities.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries on legs.
* Osteoporosis.

PD subjects:

Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Balance Performance | Baseline, 4 weeks and 8 weeks.
  Measured by the duration the stance can be maintained. Unit：seconds(s)
COP Path Length in Balance Tasks | Baseline, 4 weeks and 8 weeks.
  The total distance traveled by the COP over a specified period. Longer path lengths can indicate increased effort to maintain balance or greater instability. Unit：millimeters(mm)
COP Displacement in Balance Tasks | Baseline, 4 weeks and 8 weeks.
  Measures of COP movement in the anterior-posterior (AP) and medial-lateral (ML) directions, offering insights into the directional tendencies of balance control. Unit：millimeters(mm)
Motor Evoked Potentials (MEPs) | Baseline, 4 weeks and 8 weeks.
  MEPs are the electrical responses recorded from muscles following stimulation of the motor cortex. They reflect the efficiency of neural transmission from the cortex to the muscle. Unit：millivolts (mV)
Intracortical Facilitation (ICF) | Baseline, 4 weeks and 8 weeks.
  ICF is measured by applying a pair of TMS pulses with a short interval (e.g., 8-15 ms) where the first (subthreshold) pulse is followed by a second (suprathreshold) pulse, leading to an increased amplitude of the MEP.
Intracortical Inhibition (ICI) | Baseline, 4 weeks and 8 weeks.
  ICI is measured similarly to ICF but with a shorter inter-stimulus interval (e.g., 1-5 ms), resulting in a suppressed MEP amplitude. This suppression reflects inhibitory processes within the cortex.
Walking Speed | Baseline, 4 weeks and 8 weeks.
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 4 weeks and 8 weeks.
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline, 4 weeks and 8 weeks.
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.

SECONDARY OUTCOMES:
COP Velocity in Balance Tasks | Baseline, 4 weeks and 8 weeks.
  The speed at which the COP moves, calculated over the duration of the balance task. Higher velocities may reflect more dynamic balance adjustments or instability. Unit：millimeters per second(mm/s)
COP Area in Balance Tasks | Baseline, 4 weeks and 8 weeks.
  The area covered by the COP trajectory during the balance task, providing an estimate of the sway envelope. A larger area might indicate poorer balance control. Unit：square millimeters(mm^2)
Double Support Time | Baseline, 4 weeks and 8 weeks.
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 4 weeks and 8 weeks.
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Swing Time | Baseline, 4 weeks and 8 weeks.
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 4 weeks and 8 weeks.
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 4 weeks and 8 weeks.
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No